CLINICAL TRIAL: NCT06939764
Title: Application of the sG8 Scale in Real-World Geriatric Oncology Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Juan LI, MD, M.D., Sichuan Cancer Hospital and Research Institute
Other Study IDs: EK2025-SG8
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Solid Cancers; Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Geriatric Screening using the sG8 scale — Geriatric screening using the sG8 scale

SUMMARY:
This study is a multicenter, prospective, observational study. The study included patients aged 65 and older with solid tumors requiring systemic anti-tumor therapy. All patients underwent screening using the sG8 scale before the start of treatment, followed by routine treatment based on a plan developed through clinician decision-making. The study did not intervene in any way with the patients' diagnosis and treatment, and relevant clinical data during the treatment process were recorded accurately for follow-up patients. Study data were obtained from the electronic medical record databases and hospital information systems of multiple centers, including Sichuan Cancer Hospital. Patient clinicopathological features, pathological diagnoses, clinical stages, previous treatment histories, as well as anti-tumor treatment regimens after patient enrollment, drug dosages per cycle, treatment start times, incidence and grades of adverse events (AEs), and tumor response were extracted and collected from the medical records. All data were entered, managed, quality-controlled, exported, and analyzed through a real-world data management platform (RWDMP).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 65 years or older.
2. Patients with confirmed malignant tumors based on definitive pathological data.
3. Patients who are assessed by clinicians to have indications for systemic anti-tumor therapy.
4. Patients with a survival time greater than 12 weeks.

Exclusion Criteria:

1. Patients who do not meet the above inclusion criteria or are considered unsuitable for this study by the investigator due to other circumstances.
2. Patients who are unwilling to cooperate in completing the sG8 scale assessment.
3. Patients who do not understand the content of this study or are unwilling to participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with confirmed pathological evidence of malignant solid tumors, requiring systemic anti-tumor therapy, and aged 65 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Estimated)
Dates: Start 2025-05-16 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of unplanned treatment delays and treatment interruptions | From date receiving anti-tumor therapy after the first screening assessment until date of disease progression or death or the end of study, whichever came first, assessed up to 12 months
  The incidence of unplanned treatment delays and treatment interruptions

SECONDARY OUTCOMES:
TRAE | From date receiving anti-tumor therapy after the first screening assessment until date of disease progression or death or the end of study, whichever came first, assessed up to 12 months
  Number and percentage of patents with treatment-related adverse events assessed by CTCAE v5.0.
ORR | From date receiving anti-tumor therapy after the first screening assessment until date of disease progression or death or the end of study, whichever came first, assessed up to 12 months
  the sum percentage of participants with CR and PR assessed by RECIST v1.1 criteria every 8-12 weeks.
PFS | From date receiving anti-tumor therapy after the first screening assessment until date of disease progression or death or the end of study, whichever came first, assessed up to 12 months.
  Systemic Progression-Free Survival assessed by the investigators using RECIST V1.1.

OTHER OUTCOMES:
OS | From date receiving anti-tumor therapy after the first screening assessment until date of death or the end of study, whichever came first, assessed up to 12 months
  Overall survival